CLINICAL TRIAL: NCT06280625
Title: The Effect of the Inclusion of Soybean Flour on Glycemic Responses of Bread, Tortilla, and Arepa to Enhance Human Nutrition
Brief Title: The Effect of the Inclusion of Soybean Flour on Glycemic Responses
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We recruited and completed all 3 interventions in 10 participants for bread and 10 for tortilla, but stopped at 8 participants (instead of 10) for arepa and two of these participants only completed 2 out of 3 interventions because funding end.
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Kenneth Dallmier Consulting, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 24388
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Overweight and Obesity
Keywords: glycemic responses; insulin; satiety
MeSH Terms: conditions — Overweight; Obesity; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: People will be evaluated with a food product prepared with different % of replacement of wheat flour for soy flour. Each person will be their own control. In other words, in randomized order, they will all be assessed with the food product prepared with the regular wheat flour (either bread, tortillas or arepas) and on two other visits with different percentages of soy flour. Participants will be allowed to be assessed in more than one food product (as they wish).
Who Masked: Participant
Masking Description: Participants will be given the food product without information on whether it is prepared 100% with wheat flour or with different soy flour %.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Bread (Experimental): Bread will be prepared with 100 % of wheat flour and with some replacements by different % of soy flour (at three concentrations)
  Interventions: Other: Replacement of wheat flour by soyflour
- Tortilla (Experimental): Bread will be prepared with 100 % of wheat flour and with some replacements by different % of soy flour (at three concentrations)
  Interventions: Other: Replacement of wheat flour by soyflour
- Arepa (Experimental): Arepa will be prepared with 100 % of wheat flour and with some replacements by different % of soy flour (at three concentrations)
  Interventions: Other: Replacement of wheat flour by soyflour

INTERVENTIONS:
Other: Replacement of wheat flour by soyflour — The intervention consist in replacing a fraction of wheat flour by soyflour

SUMMARY:
Foods that release glucose rapidly, leading to spikes in blood sugar and insulin (known as high glycemic index foods), generate lower satiety responses than foods with low glycemic index. High glycemic index foods are also linked to an increased risk of developing diabetes. The partial replacement of carbohydrates in rich staple foods with soy flour has the potential to reduce glycemic response and improve satiety.

In many regions of Latin America, as well as in the Middle East and North Africa (MENA) regions, bread is the staple source of calories, but it is a relatively poor source of balanced nutrition. Bread enriched with soy flour could provide higher dietary protein while moderating blood glucose (and insulin) spikes, which can help reduce insulin resistance and metabolic diseases. The results of this study could provide government and private human nutritionists with the evidence they need to formulate soy flour into bread, corn tortillas, and arepas for schools and homes.

DETAILED DESCRIPTION:
The purpose of this study is to compare different percentages of soy flour inclusion rates in recipes of bread, flour tortilla, and arepa (South American corn pancake) for its effect on satiation and glycemic and insulin responses.

The hypothesis to be tested is that soy flour inclusion will improve the protein content, satiety profile and glycemic response of the products without significant increases in insulin responses (compared to the same products prepared with regular wheat flour).

ELIGIBILITY:
Inclusion Criteria:

* Male and female between 21-45 years of age
* All races/ethnicities
* Body mass Index (BMI) > 25 kg/m2 and <40 kg/m2 (i.e., overweight and obesity, excluding severe obesity)
* Fat %: > 30% for female or > 20% for male

Exclusion Criteria:

* Currently smokes or quit smoking nicotine cigarettes, vapes or E-cigarettes for less than 6 months ago
* Pregnant, breastfeeding, menopausal
* Hemoglobin: <11g/dl for female and <13g/dl for male
* Blood donation in the past 8 weeks
* Gluten intolerance (Gluten allergy, wheat allergy, celiac disease), Soy intolerance or allergy
* Presence of malabsorption syndrome
* History of bariatric surgery
* Presence of inflammatory intestinal disease, liver, or kidney disease
* Diabetes (fasting glucose level >126mg/dl or plasma glucose level 2h after glucose challenge >200 mg/dl) or taking medicines to treat diabetes
* Polycystic ovary syndrome (pcos)
* Untreated hypertension
* Taking any medication that might affect glucose metabolism or the results of our study
* History of cancer <5 years ago
* Abnormalities in the metabolic panel test (e.g., liver enzymes >2 times the upper limit).
* Seizures

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2024-03-11 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Plasma glucose | -30 minutes to 120 min post-prandially
  Concentrations of glucose in plasma before and at different times post-prandially
Plasma insulin | -30 minutes to 120 min post-prandially
  Concentrations of insulin in plasma before and at different times post-prandially

SECONDARY OUTCOMES:
Hunger-Satiety | Before and after (10-180 min) they consume the different food products (bread, arepa, tortillas)
  Scores in the visual analog scales assessing hunger, fullness, the prospect of eating, etc

CONTACTS AND LOCATIONS:
Overall Officials: Marta Y Pepino de Gruev, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois at Urbana Champaign, Champaign, Illinois, United States

IPD SHARING:
Plan to Share IPD: No